CLINICAL TRIAL: NCT00941967
Title: Randomized Phase II Trial Assessing the Combination of Nexavar® (Sorafenib), and Gemcitabine/Oxaliplatin in Patients Treated for Advanced (Unresectable/Metastatic) Hepatocellular Carcinoma.
Brief Title: Sorafenib With or Without Gemcitabine and Oxaliplatin in Treating Patients With Locally Advanced, Unresectable, or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CDR0000638394; CLCC-GONEXT-PRODIGE-10; VA 2007/40; INCA-RECF0917; EUDRACT-2008-000123-26
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2017-08

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; advanced adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Gemcitabine; Oxaliplatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive oral sorafenib tosylate as in arm I. Patients also receive gemcitabine hydrochloride IV over 100 minutes on day 1 and oxaliplatin IV over 2 hours on day 2. Treatment with gemcitabine hydrochloride and oxaliplatin repeats every 14 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate
- Arm II (Experimental): Patients receive oral sorafenib tosylate twice daily on days 1-14.
  Interventions: Drug: gemcitabine hydrochloride; Drug: oxaliplatin; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Arms: Arm II
Drug: oxaliplatin — Given IV
  Arms: Arm II
Drug: sorafenib tosylate — Given orally.

SUMMARY:
RATIONALE: Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as gemcitabine hydrochloride and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether sorafenib tosylate is more effective when given with or without gemcitabine hydrochloride and oxaliplatin in treating patients with liver cancer.

PURPOSE: This randomized phase II trial is studying sorafenib tosylate to see how well it works when given with or without gemcitabine hydrochloride and oxaliplatin in treating patients with locally advanced, unresectable, or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess progression-free survival (RECIST) in patients with locally advanced, unresectable or metastatic hepatocellular carcinoma treated with sorafenib tosylate with vs without gemcitabine hydrochloride and oxaliplatin.

Secondary

* Evaluate the tolerability of these regimens in these patients.
* Determine the objective response rate (RECIST) in patients treated with these regimens.
* Assess the overall survival of patients treated with these regimens.
* Evaluate the pharmacokinetics of sorafenib tosylate.
* Assess biomarkers (e.g., pERK levels) associated with treatment response.
* Assess angiogenic response by functional imaging.

OUTLINE: This is a multicenter study. Patients are stratified according to performance status and CLIP score. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sorafenib tosylate as in arm I. Patients also receive gemcitabine hydrochloride IV over 100 minutes on day 1 and oxaliplatin IV over 2 hours on day 2. Treatment with gemcitabine hydrochloride and oxaliplatin repeats every 14 days for 12 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral sorafenib tosylate twice daily on days 1-14. In both arms, courses with sorafenib tosylate repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Blood samples and/ or tumor tissue samples may be collected for further analysis.

After completion of study therapy, patients are followed every 2 months until disease progression and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma not amenable to liver transplantation

  * Locally advanced, unresectable, or metastatic disease
* At least 1 lesion accurately measured in ≥ 1 dimension according to RECIST criteria AND has not been previously treated with local therapy (e.g., intra-arterial chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation)

  * No presence of bone metastasis only
* No known brain metastasis

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy > 12 weeks
* ANC > 1,500/mm^3
* WBC > 3,000/mm^3
* Platelet count ≥ 90,000/mm^3
* Hemoglobin > 10 g/dL
* Total protein ≥ 40%
* ALT or AST ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* Amylase and lipase < 1.5 times ULN
* Creatinine < 1.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* Albumin ≥ 2.8 mg/dL
* INR ≤ 2.3
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study and for up to 4 months for females and 6 months for males after completion of study treatment
* CLIP score 0-3
* No Child Pugh score B or C cirrhosis
* No known HIV positivity
* No other prior malignancy, except adequately treated or curative basal cell skin cancer or carcinoma in situ of the cervix
* No known or suspected allergy to the investigational agent or any agent given in association with this study
* No cardiovascular disease, including any of the following:

  * Cardiac arrhythmia requiring antiarrhythmic therapy, except beta-blockers or digoxin for chronic atrial fibrillation
  * Active coronary artery disease or ischemia
  * Myocardial infarction within the past 6 months
  * NYHA class II-IV congestive heart failure
* No uncontrolled hypertension
* No severe active bacterial or fungal infection > CTCAE v3.0 grade 2
* No peripheral neuropathy ≥ grade 2
* No condition that could affect the absorption of study drug, including any of the following:

  * Malabsorption syndrome
  * Disease significantly affecting gastrointestinal function
  * Bowel obstruction or sub-obstruction
* No dysphagia or inability to swallow tablets
* No history of seizures requiring long-term antiepileptic treatment
* No unstable condition that would jeopardize safety or compliance with study including any of the following :

  * Medical, psychological, or social conditions
  * Substance abuse
  * Legal incapacity or limited legal capacity
* No psychological, familial, social, or geographic reasons that would preclude clinical follow-up
* Must be registered in a social security program

PRIOR CONCURRENT THERAPY:

* No prior organ transplantation with immunosuppressive treatment
* No prior systemic chemotherapy or systemic antiangiogenic treatment for hepatocellular carcinoma
* No prior major resection of the stomach or proximal small bowel
* Prior anticoagulation therapy (e.g., warfarin or heparin) allowed with INR parameters within normal limit range
* At least 4 weeks since prior local therapy to lesions and treated lesions may not be selected as target lesions
* No concurrent or prior long-term treatment with CYP3A4 inducers (e.g., rifampin, hypericum perforatum, phenytoin, carbamazepine, phenobarbital, and dexamethasone)
* No concurrent antitumoral treatment, including tamoxifen, interferon, or somatostatin analogues
* No other concurrent experimental drugs or anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tumor response according to RECIST criteria | 18 months
Progression-free survival | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Assenat, MD, Principal Investigator — Hopital Saint Eloi
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Blay JY, Bonvalot S, Casali P, Choi H, Debiec-Richter M, Dei Tos AP, Emile JF, Gronchi A, Hogendoorn PC, Joensuu H, Le Cesne A, McClure J, Maurel J, Nupponen N, Ray-Coquard I, Reichardt P, Sciot R, Stroobants S, van Glabbeke M, van Oosterom A, Demetri GD; GIST consensus meeting panelists. Consensus meeting for the management of gastrointestinal stromal tumors. Report of the GIST Consensus Conference of 20-21 March 2004, under the auspices of ESMO. Ann Oncol. 2005 Apr;16(4):566-78. doi: 10.1093/annonc/mdi127. PMID 15781488
- [Background] Blay JY, Landi B, Bonvalot S, Monges G, Ray-Coquard I, Duffaud F, Bui NB, Bugat R, Chayvialle JA, Rougier P, Bouche O, Bonichon F, Lassau N, Vanel D, Nordlinger B, Stoeckle E, Meeus P, Coindre JM, Scoazec JY, Emile JF, Ranchere D, Le Cesne A. [Recommendations for the management of GIST patients]. Bull Cancer. 2005 Oct;92(10):907-18. French. PMID 16266874
- [Background] Lassau N, Lamuraglia M, Leclere J, Rouffiac V. [Functional and early evaluation of treatments in oncology: interest of ultrasonographic contrast agents]. J Radiol. 2004 May;85(5 Pt 2):704-12. doi: 10.1016/s0221-0363(04)97651-2. French. PMID 15238871
- [Background] Lassau N, Chami L, Peronneau P. [Current events about echography in 2006: position of the ultrasound functional imaging for the early evaluation of targeted therapeutics]. Bull Cancer. 2006 Dec;93(12):1207-11. French. PMID 17182377
- [Background] Lassau N, Lamuraglia M, Chami L, Leclere J, Bonvalot S, Terrier P, Roche A, Le Cesne A. Gastrointestinal stromal tumors treated with imatinib: monitoring response with contrast-enhanced sonography. AJR Am J Roentgenol. 2006 Nov;187(5):1267-73. doi: 10.2214/AJR.05.1192. PMID 17056915
- [Background] Lamuraglia M, Escudier B, Chami L, Schwartz B, Leclere J, Roche A, Lassau N. To predict progression-free survival and overall survival in metastatic renal cancer treated with sorafenib: pilot study using dynamic contrast-enhanced Doppler ultrasound. Eur J Cancer. 2006 Oct;42(15):2472-9. doi: 10.1016/j.ejca.2006.04.023. Epub 2006 Sep 11. PMID 16965911
- [Background] Escudier B, Lassau N, Angevin E, Soria JC, Chami L, Lamuraglia M, Zafarana E, Landreau V, Schwartz B, Brendel E, Armand JP, Robert C. Phase I trial of sorafenib in combination with IFN alpha-2a in patients with unresectable and/or metastatic renal cell carcinoma or malignant melanoma. Clin Cancer Res. 2007 Mar 15;13(6):1801-9. doi: 10.1158/1078-0432.CCR-06-1432. PMID 17363536